CLINICAL TRIAL: NCT05097651
Title: Pilot Trial of Cannabidiol (CBD) for Sleep Problems in People With HIV
Brief Title: CBD for Sleep in People With HIV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties enrolling eligible participants
Sponsor: Mariana Cherner, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Mariana Cherner, PhD, Professor IR, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201536; R21DA053160 (NIH)
Record Dates: First submitted 2021-10-05; First posted 2021-10-28 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD (Experimental): Participants will receive oral liquid cannabidiol
  Interventions: Drug: Cannabidiol oral solution
- Placebo (Placebo Comparator): Participants will receive an inert oral liquid
  Interventions: Drug: Inert sesame seed oil

INTERVENTIONS:
Drug: Cannabidiol oral solution — Cannabidiol 100mg/mL in a sesame seed oil, strawberry flavored solution, taken orally at bedtime in self-titrated dose between 50mg and 600mg. Once a dose that results in relief of symptoms is reached, it will remain as the maintenance dose, not to exceed 600mg.
  Arms: CBD
Drug: Inert sesame seed oil — Placebo will be identical strawberry flavored sesame seed oil-based solution without CBD.
  Arms: Placebo

SUMMARY:
This study will obtain preliminary information about whether, and at what dose, cannabidiol (CBD) may help with insomnia in people living with human immunodeficiency virus (HIV). The study will be a 5-week randomized, double-blind placebo-controlled phase II trial using daily oral CBD doses between 50mg and 600mg. Sleep problems will be measured using a wrist-worn device and by self-report. Performance on tests of thinking skills will be compared before and after CBD/placebo treatment. Positive study results will provide support for the use of CBD as a potential treatment for insomnia.

DETAILED DESCRIPTION:
Sleep problems are highly prevalent in people with HIV, and traditional treatment with sedative/hypnotic medications can compound neurocognitive dysfunction. A treatment option without cognitive side effects would be highly desirable for use with this vulnerable population. Cannabidiol (CBD) is a phytocannabinoid component of the marijuana plant that is considered devoid of euphoriant or other psychoactive properties. A small literature demonstrates a broad range of CBD doses at which sleepiness is reported to occur, and also not occur, which indicates the need for controlled studies to ascertain the lowest efficacious dose, as well as the sustainability of effects over a period of repeated use. The proposed clinical trial will seek to 1) Ascertain the dose range of CBD that is useful in managing symptoms of insomnia and improving sleep quality, and 2) determine whether CBD use has any next-morning cognitive sequelae measured objectively with a neuropsychological test battery.

In the proposed five-week clinical trial, investigators will use a liquid solution that is 100 mg/mL of CBD formed from semi synthetic CBD powder suspended in sesame oil. Eligible participants will be randomized into either a CBD or Placebo group. At the baseline visit, participants will be fitted with a wrist-worn actigraph to measure activity and light exposure, which they were wear for 5 weeks to estimate their rest/ activity cycle.

After a 7-day baseline period, participants will be instructed to take 50mg of CBD/placebo to begin the titration phase. They will slowly increase their daily dose by 100mg/day until they achieve relief from symptoms of insomnia. This includes the option to remain on the minimum study dose of 50 mg daily to a maximum medication limit of 600 mg daily. Participants will return weekly to monitor vital signs, download actigraphy data, and receive the next allotment of study medication. Clinical labs, self-reported sleep, fatigue, and mood, as well neuropsychological test performance will be be measured at baseline and at the end of the medication maintenance phase. Participants will also be instructed to use a daily diary to record sleep and other health related items, as well as adherence to the study regimen for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ and HIV- adults with complaints of sleep problems
* Ability to provide informed consent;
* Read, speak, and understand English or Spanish as a first language;
* Willingness to stop sedative/hypnotic medication use;
* Willingness to abstain from substance use;
* Willingness to prevent pregnancy.

Exclusion Criteria:

* Inability to provide informed consent;
* Medical conditions other than HIV disease that may confound study results or pose risk when participating in the study;
* Neurologic disorder that could compromise interpretation of study findings, such as seizure disorder, stroke, demyelinating diseases, or head injury with loss of consciousness for greater than 30 minutes or resulting in neurologic complications; and other non-HIV neurological disorders;
* Severe psychiatric disorder that might make the person's participation in the study problematic or unsafe, including psychiatric disorder with psychotic features, severe depression, or suicidality;
* Current sedative/hypnotic use for a non-sleep related indication or abuse within the last 12 months;
* Use of marijuana, CBD, or other natural or synthetic cannabinoids in the last 30 days;
* Any moderate to severe substance use disorder (dependence) in the last 12 months;
* Any mild substance use disorder (abuse) in the last 30 days;
* Pregnancy or lactation, or unwillingness to prevent pregnancy during the trial;
* Compromised liver or kidney function;
* Evidence of cardiovascular risk,
* Uncontrolled hypertension;
* Chronic pulmonary disease;
* Obstructive sleep apnea, narcolepsy, or other non-insomnia sleep diagnosis;
* Overnight-shift work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in sleep latency assessed by wrist-worn actigraphy | At baseline before treatment and after completion of the medication phase at 4 weeks
  We will determine whether the study drug affects how quickly people fall asleep using a motion/activity sensor called an actigraph that is worn on the wrist.

SECONDARY OUTCOMES:
Change in sleep quality assessed by the Pittsburgh Sleep Quality Index | At baseline before treatment and after completion of the medication phase at 4 weeks
  We will determine whether the study drug affects self-reported sleep quality using a paper-and-pencil measure called the Pittsburgh Sleep Quality Index. Scores can range from 0 to 21, with higher score indicating more sleep problems.
Change in neurocognitive function based on a combination of tests that measure thinking skills | At baseline before treatment and after completion of the medication phase at 4 weeks
  Change in a summary score based on a combination of demographically adjusted neuropsychological tests with known sensitivity to effects of HIV and the Fluid Composite T-score on the Cognition module of the NIH Toolbox for the Assessment of Neurological and Behavioral Function. T-scores can range between 1-100, with higher scores reflecting better performance

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Cherner, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego School of Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and biospecimens collected in the course of this study will be stored in the joint HIV Neurobehavioral Research Center (HNRP) - Center for Medicinal Cannabis Research (CMCR) Data and Biospecimen Repositories for potential future use. De-identified data and biospecimens may be made available to investigators conducting institutional review board (IRB) approved research. Interested investigators will submit a request for data and/or biospecimens. HNRP-CMCR leadership will be responsible for determining who will have access to the data and biospecimens and will ensure that a Data Use Agreement is signed by the requesting investigator. The data and biospecimens will be stored indefinitely, however, if a research participant decides they no longer want their biospecimens to be used, all efforts will be made to stop any additional studies.
Time Frame: The data and biospecimens will become available following publication. Data and biospecimens will be stored indefinitely, however, if a research participant decides they no longer want their biospecimens to be used, all efforts will be made to stop any additional studies.
Access Criteria: Investigators whose proposed use of the data and/or biospecimens has been approved by the HNRP-CMCR leadership. HNRP-CMCR leadership will ensure that a Data Use Agreement is signed by the requesting investigator.
URL: https://www.cmcr.ucsd.edu/